CLINICAL TRIAL: NCT07254793
Title: A Feasibility/Pilot First-in-human Study of Exercise-mobilized NK-enriched Donor Lymphocyte Infusions (DLI-X) to Prevent or Treat Leukemia Relapse After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Prophylactic and Therapeutic DLI-X for Leukemia Relapse After HCT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006003
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoid Leukemia; Acute Myeloid Leukemia; Acute Undifferentiated Leukemia (AUL); Myelodysplastic Syndrome; Chronic Myeloid Leukemia; Non-Hodgkin Lymphoma
Keywords: Exercise; Donor Lymphocyte Infusion; Allogeneic Hematopoietic Stem Cell Transplantation; Hematologic Malignancies; Matched Sibling Donor; Haploidentical; Hematopoietic Cell Transplantation; DLI-X
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Motor Activity; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prophylactic Arm (Experimental): Conduct the first-in-human, randomized clinical trial comparing prophylactic exercise mobilized donor lymphocyte infusion (pro-DLI-X) with standard (non exercise mobilized) prophylactic DLI (pro-DLI) for relapse prevention following allogeneic hematopoietic cell transplantation (alloHCT) in patients with myeloid or lymphoid malignancies.
  Interventions: Biological: Exercise Mobilized Prophylactic DLI; Biological: Standard Prophylactic DLI
- Therapeutic Arm (Experimental): Compare therapeutic exercise mobilized donor lymphocyte infusion (t-DLI-X) with standard (non exercise mobilized) therapeutic DLI (t-DLI) in a randomized trial for patients with evidence of minimal residual disease (MRD+) or overt relapse post-alloHCT for myeloid or CD19-negative lymphoid malignancies.
  Interventions: Biological: Exercise Mobilized Therapeutic DLI; Biological: Standard Therapeutic DLI

INTERVENTIONS:
Biological: Exercise Mobilized Prophylactic DLI — Pro-DLI-X will be given through the patient's central line at an initial dose of 100,000 CD3+ cells/kilogram (kg) of recipient weight for haploidentical hematopoietic cell transplantation (haploHCT) and 300,000 CD3+ cells/kg for matched sibling donor hematopoietic cell transplantation (MSD HCT). Participants will receive up to 3 doses of pro-DLI-X, and each dose will be increased as follows: dose 2 will be 300,000 CD3+ cells/kg for haploHCT and 1,000,000 CD3+ cells/kg for MSD HCT; dose 3 will be 1,000,000 CD3+ cells/kg for haploHCT and 3,000,000 CD3+ cells/kg for MSD HCT.
  Other Names: pro-DLI-X
  Arms: Prophylactic Arm
Biological: Standard Prophylactic DLI — Pro-DLI will be given through the patient's central line at an initial dose of 100,000 CD3+ cells/kilogram (kg) of recipient weight for haploidentical hematopoietic cell transplantation (haploHCT) and 300,000 CD3+ cells/kg for matched sibling donor hematopoietic cell transplantation (MSD HCT). Participants will receive up to 3 doses of pro-DLI-X, and each dose will be increased as follows: dose 2 will be 300,000 CD3+ cells/kg for haploHCT and 1,000,000 CD3+ cells/kg for MSD HCT; dose 3 will be 1,000,000 CD3+ cells/kg for haploHCT and 3,000,000 CD3+ cells/kg for MSD HCT.
  Other Names: pro-DLI
  Arms: Prophylactic Arm
Biological: Exercise Mobilized Therapeutic DLI — t-DLI-X will be given through the patient's central line at an initial dose of 1,000,000 CD3+ cells/kilogram (kg) of recipient weight for haploidentical hematopoietic cell transplantation (haploHCT) and 3,000,000 CD3+ cells/kg for matched sibling donor hematopoietic cell transplantation (MSD HCT). Participants will receive up to 3 doses of t-DLI-X, and each dose will be increased as follows: dose 2 will be 3,000,000 CD3+ cells/kg for haploHCT and 10,000,000 CD3+ cells/kg for MSD HCT; dose 3 will be 10,000,000 CD3+ cells/kg for haploHCT and 30,000,000 CD3+ cells/kg for MSD HCT.
  Other Names: t-DLI-X
  Arms: Therapeutic Arm
Biological: Standard Therapeutic DLI — t-DLI will be given through the patient's central line at an initial dose of 1,000,000 CD3+ cells/kilogram (kg) of recipient weight for haploidentical hematopoietic cell transplantation (haploHCT) and 3,000,000 CD3+ cells/kg for matched sibling donor hematopoietic cell transplantation (MSD HCT). Participants will receive up to 3 doses of t-DLI-X, and each dose will be increased as follows: dose 2 will be 3,000,000 CD3+ cells/kg for haploHCT and 10,000,000 CD3+ cells/kg for MSD HCT; dose 3 will be 10,000,000 CD3+ cells/kg for haploHCT and 30,000,000 CD3+ cells/kg for MSD HCT.
  Arms: Therapeutic Arm

SUMMARY:
The primary objective of this proposal is to conduct the first-in-human randomized clinical trial evaluating prophylactic DLI-X (pro-DLI-X) for relapse prevention following matched sibling donor (MSD) or haploidentical (haplo) hematopoietic cell transplantation (HCT) in patients with hematologic malignancies. Additionally, the study aims to assess the safety and efficacy of therapeutic DLI-X (t-DLI-X) compared to t-DLI alone in patients with minimal residual disease (MRD+) or overt relapse post-alloHCT. For patients with CD19-positive lymphoid malignancies, the study will incorporate blinatumomab, while those with myeloid or CD19-negative lymphoid malignancies will receive t-DLI-X or t-DLI alone.

We hypothesize that both pro-DLI-X and t-DLI-X, with or without blinatumomab, will demonstrate safety and superior efficacy by enhancing graft-versus-leukemia (GvL) effects mediated by natural killer (NK) cells, γδ T cells, and CD8+ T cells, while maintaining manageable and treatment-responsive graft-versus-host disease (GvHD).

ELIGIBILITY:
DLI Recipient Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 0-65 years
* Diagnosis of acute leukemia (lymphoid, myeloid or undifferentiated) myelodysplastic syndrome (MDS), chronic myeloid leukemia (CML) or non-Hodgkin's lymphoma (NHL)
* Undergoing myeloablative or reduced intensity matched sibling donor (MSD) HCT or haploidentical HCT
* Have a locally available healthy matched or haploidentical (≥5/10 HLA antigen matched) related donor between 12 and 50 years of age, consented and able to perform the exercise sessions. (see donor inclusion criteria)
* The familial donors will first complete the fitness evaluation to determine VO2max and peak cycling power and following successful completion of the donor evaluation, the patients willing to participate in the randomized trial will be enrolled.

DLI Donor Inclusion Criteria:

* Matched sibling donor or HLA-haploidentical relatives of the patient, including biological parents, siblings, or children, half-siblings, cousins or aunts and uncles
* Weight is greater than 30 kg
* Age 12 and 50 years
* Ability to undergo phlebotomy
* Cardiac, renal, pulmonary, and hepatic function within normal limits
* Complete blood count (CBC) with differential and platelet count within normal limits, and CMP within normal limits as deemed acceptable by the Principal Investigator and provider evaluating donor.
* The familial donors should be able complete the fitness evaluation to determine VO2max and peak cycling power and following successful completion of the donor evaluation, the patients willing to participate in the randomized trial will be enrolled.

DLI Recipient Exclusion Criteria:

* Acute grade III-IV aGvHD or moderate/severe chronic GvHD.
* Requiring immunosuppression therapy for treatment of GvHD.
* Co-morbidities: AST/ALT greater than 5 x ULN; Bilirubin greater than 2 x ULN; Creatinine greater than 2 x ULN for age or creatinine clearance/GFR <40 ml/min/1.73m2; Pulmonary function: DLCO less than 40% of normal or O2 Sat less than 92%; Cardiac: left ventricular ejection fraction less than 35%; active infection; HIV positive; Karnofsky score (adults) less than 60% or Lansky score less than 50% (pediatrics)
* Uncontrolled or severe bacterial, fungal or viral infection.
* Positive serum or urine pregnancy test for girls post menarche or women of childbearing age.
* Severe psychiatric illness or mental deficiency making compliance to treatment unlikely and/or informed consent impossible.
* Any reason, at the investigator's discretion, that the participation of the patient in this protocol would not be in patient's best interest, or where the patient would be unable to adhere to the study requirements.

DLI Donor Exclusion Criteria:

* Unable to perform graded exercise test
* Cardiac or pulmonary disease restricting exercise
* Positive anti-donor HLA antibody
* Pregnant or lactating
* Active infection
* Positivity for HIV, hepatitis B (HBV), hepatitis C (HCV), human T-cell lymphotropic virus (HTLV-I/II)
* Severe psychiatric illness or mental deficiency making compliance with donation unlikely and/or informed consent impossible.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Prophylactic endpoint: Graft-versus-Host Disease-Free, Relapse-Free Survival (GRFS) | Assess between 1 to 3 years post HCT
  Graft-versus-Host Disease-Free, Relapse-Free Survival (GRFS) is defined as survival without evidence of disease relapse or grade III-IV acute graft-versus-host-disease (aGvHD) or chronic graft-versus-host-disease (cGvHD) requiring systemic therapy. In essence, GRFS serves as a meaningful measure encompassing not only survival but quality of life. GRFS will be compared in patients randomized to pro-DLI-X versus standard pro-DLI control group.
Therapeutic endpoint: Disease response to t-DLI versus t-DLI-X (relapse and GvHD rates as a composite endpoint) | Assess between 1-3 years post HCT
  A parallel two-group design will be used to test whether the percent response to t-DLI-X (treatment) is different from the percent response to t-DLI (control).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Katsanis, MD, Principal Investigator — University of Arizona
Locations (1):
- The University of Arizona Cancer Center, Tucson, Arizona, United States